CLINICAL TRIAL: NCT03814057
Title: Age- Adjusted Measurements of Creatinine Height Index for Diagnosing Malnutrition in Elderly Medical Patients at Hospital Admission
Brief Title: Creatinine Height Index in Elderly
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doha Rasheedy, Assistant Professor of Geriatric Medicine, Ain Shams University
Other Study IDs: AinShamsGer
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Malnutrition in Elderly
Keywords: Anthropometric measurements,; creatinine height index; lean body mass; Mini- nutritional assessment; Hand Grip strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Medical Patients at hospital admission
  Interventions: Diagnostic Test: 24 hour urine creatinine excretion

INTERVENTIONS:
Diagnostic Test: 24 hour urine creatinine excretion — two age corrected calculations of creatinine height index were obtained

SUMMARY:
evaluation of the efficacy of two different age adjusted calculations of CHI compared to other nutritional indicators in the elderly medical patients upon hospital admission.

DETAILED DESCRIPTION:
Cross sectional study involving one hundred hospitalized elderly (>60 years), Anthropometric measurements, Mini- nutritional assessment, Hand Grip strength, CBC, total protein, albumin, total cholesterol, triglyceride, and 24 hour urinary creatinine excretion were measured within 24 hours of hospital admission calculation of CHI using 2 age adjusted modification was done accuracy of each measurement in detecting malnutrition was evaluated

ELIGIBILITY:
Inclusion Criteria:

* medical elderly patients (>60 years)
* within 24 hours of hospital admission

Exclusion Criteria:

* sepsis
* fever
* malignancy
* liver cirrhosis
* renal impairment
* critically ill patients
* those with any hemodynamic instability were excluded from the study
* patients receiving diuretics
* patients can't stand to obtain their weight and height
* those can't collect 24 hour urine
* the patients refused to participate in the study

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly Medical Patients at hospital admission with exclusion of factors might affect 24 hour urine collection or urinary creatinine excretion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
accuracy of creatinine height index in Elderly | within 24 hours of hospital admission
  evaluate the test performance of the two age adjusted calculations of creatinine height index for detecting malnutrition in elderly patients at hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: DOHA RASHEEDY, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt